CLINICAL TRIAL: NCT00731900
Title: Pharmacogenetic Study for Topiramate-Induced Cognitive Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Hrong-Huei Liou, MD;PhD, National Taiwan University Hospital
Other Study IDs: 9561707009
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-08

CONDITIONS: Cognitive Dysfunction
Keywords: pharmacogenetic; study; Topirmate; induced
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Topiramate (TPM) is an antiepileptic drug with a unique mode of action that is often useful in patients refractory to other drugs. However its use is restricted by the high incidence of cognitive adverse drug reactions (ADRs) that are associated with TPM exposure. TPM has been shown to cause particular cognitive ADRs, characterized by verbal fluency, attention, working memory and language deficits, at a much higher rate than other antiepileptic drugs. There do not appear to be obvious differences between patients that do or do not experience cognitive ADRs when on TPM (e.g. age, sex, concomitant medications, diagnosis), which suggests a genetic contributor.

ELIGIBILITY:
Inclusion Criteria:

* adult (>17 years old) patients with epilepsy or patients with migraine treated by topiramate

Exclusion Criteria:

* allergy to topiramate
* abnormal liver or renal function

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with epilepsy or patients with migraine treated by topiramate
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Horng-Huei Liou, MD;PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan